CLINICAL TRIAL: NCT07396298
Title: The Effects and Mediating Mechanism of the Existential Cognitive Intervention to Enhance Positive Aspect of Caregiving (EXCITE-PAC) in a Dementia Context: A Sequential Mixed Method Study
Brief Title: The Existential Cognitive Intervention to Enhance Positive Aspect of Caregiving (EXCITE-PAC) in a Dementia Context
Acronym: EXCITE-PAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Proferssor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXCITE-PAC
Record Dates: First submitted 2025-12-14; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dementia Caregiver
Keywords: Positive aspect of caregiving; dementia caregiver; existential-cognitive intervention

STUDY DESIGN:
Intervention Model Description: The EXCITE-PAC program is an overall 12-week training and comprises of three phases as follows:
  1. Face-to-face home visit (week 1) - it will commence with a home visit to establish narrative-based caregiver biographies.
  2. Group-based virtual meetings (Weeks 2-8), Over the next 7 weeks, weekly virtual group-based meetings will be held during which video-guided self-distancing cognitive reappraisal will be used to enhance emotional regulation and meaning-making. The goal-oriented empowerment approach will be used in the virtual meetings to facilitate carers' use of reframing and refocusing techniques in the day-to-day caregiving process to promote the evolvement of PAC.
  3. telephone follow-ups (Weeks 10-12) - Thereafter, two bi-weekly telephone calls will be made to continue supporting goal attainment.
Who Masked: Outcomes Assessor
Masking Description: The pilot randomized controlled trial will be conducted in two elderly community centers of a non-government organization in Hong Kong. Participants will be randomized into intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : EXCITE-PAC program (Experimental): The EXCITE-PAC program is an overall 12-week training and comprises of three phases as follows:
  1. Face-to-face home visit (week 1) - it will commence with a home visit to establish narrative-based caregiver biographies.
  2. Group-based virtual meetings (Weeks 2-8), Over the next 7 weeks, weekly virtual group-based meetings will be held during which video-guided self-distancing cognitive reappraisal will be used to enhance emotional regulation and meaning-making. The goal-oriented empowerment approach will be used in the virtual meetings to facilitate carers' use of reframing and refocusing techniques in the day-to-day caregiving process to promote the evolvement of PAC.
  3. telephone follow-ups (Weeks 10-12) - Thereafter, two bi-weekly telephone calls will be made to continue supporting goal attainment.
  Interventions: Other: existential-cognitive intervention to enhance PAC
- Usual care (Placebo Comparator): Usual care will be provided to the control group which mainly covers the social activities offered by the affiliated center. The participants are requested not to join any activities relating to cognitive training or auditory training before the post-test data collection.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: existential-cognitive intervention to enhance PAC — The EXCITE-PAC program is an overall 12-week training and comprises of three phases as follows:
  1. Face-to-face home visit (week 1) - it will commence with a home visit to establish narrative-based caregiver biographies.
  2. Group-based virtual meetings (Weeks 2-8), Over the next 7 weeks, weekly virtual group-based meetings will be held during which video-guided self-distancing cognitive reappraisal will be used to enhance emotional regulation and meaning-making. The goal-oriented empowerment approach will be used in the virtual meetings to facilitate carers' use of reframing and refocusing techniques in the day-to-day caregiving process to promote the evolvement of PAC.
  3. telephone follow-ups (Weeks 10-12) - Thereafter, two bi-weekly telephone calls will be made to continue supporting goal attainment.
  Arms: Experimental : EXCITE-PAC program
Other: Usual care — Usual care will be provided to the control group which mainly covers the social activities offered by the affiliated center. The participants are requested not to join any activities relating to cognitive training or auditory training before the post-test data collection.
  Arms: Usual care

SUMMARY:
Although research evidence is emerging on the co-existence of a positive caregiving experience in the physically and psychosocially taxing dementia care context, little attention has been paid to promoting the positive aspects of caregiving (PAC) among family carers. We adopt the paradigm of existential positive psychology, integrating cognitive behavioural theory, construal level theory, and Antonovsky's theory of salutogenesis to develop an existential-cognitive intervention to enhance positive aspects of caregiving (EXCITE-PAC), and thereby improve the health outcomes of family carers of people living with dementia (PLwD). A randomised controlled trial is proposed to evaluate the effects of EXCITE-PAC on carers' health and to examine whether any such effects are mediated through changes in PAC. Post-trial interviews with carers will further elucidate their experiences of the intervention and their perceptions of its impact.

The proposed study will yield important theoretical and public health advances. Theoretically, it will test the validity of an integrative paradigm designed to enrich the life space of family carers in the context of dementia care by increasing their opportunities to experience PAC. If supported, this paradigm can complement the dominant stress-coping framework and help reshape the caregiving experience of family carers of PLwD. From a public health perspective, if EXCITE-PAC proves effective, it will respond to the WHO Global Action Plan on Dementia by promoting carers' health. Crucially, by enriching carers' PAC through empowering them to internalise a new perspective on dementia caregiving, the intervention has the potential to foster more sustainable and evolving positive effects on role adaptation and health status. Together with a comprehensive evaluation of outcomes and end-user experiences, the knowledge generated from this study can be readily translated into dementia care service development and policy. This is a pilot mixed-method study comprising a randomised controlled trial and a post-trial qualitative interview. The inclusion criteria are: i) family carers of Chinese PLwDs diagnosed at least six months previously; ii) caregiving for ≥ 4 hours/day; iii) Chinese-speaking; iv) have a mobile device to access virtual meetings via Go-To-Meeting or Zoom; and iv) consent to participate. After the baseline outcome evaluation, they will be randomised to receive the 12-week EXCITE-PAC program or usual care. The program comprises three phases, including i) face-to-face home visit, ii) group-based virtual meetings, and iii) telephone follow-ups. The outcome evaluation on i) PAC, ii) Health-related quality of life (HRQoL), iii) depression, iv) self-efficacy in caregiving, and v) meaning-making upon programme completion will be assessed at baseline, in the 12th and 18th weeks. Qualitative interviews will be conducted.

DETAILED DESCRIPTION:
The global prevalence of dementia is escalating. Alzheimer's Disease International reports that 10 million people worldwide are diagnosed with dementia each year, indicating that there will be 78 million people living with dementia (PLwD) by 2030 and 139 million by 2050. The economic implications are significant, with the global cost of care estimated to total US$2 trillion by 2030. Figures from 2019 suggest that about 50% of this cost can be attributed to informal care, the majority of it provided by family caregivers. Supporting family carers of PLwD has therefore been recognised by the World Health Organisation as a high priority in the Global Action Plan on Dementia 2017-2025.

As a progressive debilitating syndrome characterised by cognitive deficits, mood and behavioural problems, and subsequent disability, dementia makes family caregiving for PLwD highly challenging, stressful and frustrating. A nationwide study on the health impact of family caregiving for PLwD found that family carers reported poorer health-related quality of life in the aspects of mobility, self-care, activity, pain/discomfort and emotions than non-carers, with the disparity remaining significant after three years. Sustaining invaluable informal care support for PLwD thus demands effective strategies for enhancing carers' role adaptation and health status.

Mainstream research on the adaptation process of family carers focuses on reducing their stressful caregiving experience and the associated health threats. Although research evidence is emerging on the co-existence of a positive caregiving experience in the physically and psychosocially taxing dementia care context, little attention has been paid to promoting the positive aspects of caregiving (PAC) among family carers. PAC is conceptualised as the extent to which the caregiving experience is seen as enriching an individual's life space and yielding positive consequences. Instead of being located at the opposite end of a caregiving burden continuum, PAC is a separate dimension that captures the experience of carers. A significant body of research has accumulated on the protective effects of PAC against the detrimental health impact of caregiving among family carers of PLwD, including lessening anxiety and depression, reducing the perceived disturbance of behavioural symptoms, and enhancing subjective health. A high level of PAC among family carers is also associated with a reduced risk of PLwD institutionalisation. The lack of a proactive method to enhance PAC for carers may be related to PAC being cultivated internally among family carers through a complex process of adjusting values and reframing the caregiving experience to schemata that are compatible with carers' own life philosophies, missions and priorities. Theoretical guidance on the evolving PAC process is therefore warranted to inform the development of interventions to promote PAC.

The investigators have developed an integrative theoretical model based on the stress coping paradigm and existential paradigm to predict PAC in the dementia context. Empirical evaluation of the model in a longitudinal cohort study elucidated the underlying mechanism explaining such evolvement. Based on these findings, the investigators adopt the paradigm of existential positive psychology, which integrates cognitive behavioural theory, construal level theory and Antonovsky's theory of salutogenesis, to pioneer an existential-cognitive intervention to enhance PAC (EXCITE-PAC), and therefore the health outcomes of family carers of PLwD. A randomised controlled trial is proposed to evaluate the effects of EXCITE-PAC on carers' health and to explore whether those effects (if any) are mediated through a change in PAC. Post-trial interviews with carers will elucidate the experience and perceived effects.

The proposed study will bring about important theoretical and public health advances. Theoretically, the study will inform the validity of an integrative theoretical paradigm to enrich the life space of family carers in the dementia care context by increasing the carer's encounters with PAC. This theoretical paradigm, if valid, can complement the stress coping paradigm to reshape the caregiving experience of family carers of PLwD. As for the public health implications, EXCITE-PAC, if proved effective, will respond to the Global Action Plan on Dementia by promoting carers' health. More importantly, as enriching the PAC of carers involves empowering them to internalise a new perspective on the experience of dementia caregiving, a more sustainable and ever-evolving positive effect on their role adaptation and health status can be expected. Together with a comprehensive evaluation of outcomes and end-users' experience, the knowledge generated from this study can be readily translated into dementia care service development and policy settings.

Overall aim & objectives

This sequential mixed-method study aims to:

i) evaluate the effects of the 12-week EXCITE-PAC programme on PAC (primary outcome), Health-related quality of life (HRQoL), depression, caregiving self-efficacy and meaning-making among the family carers of PLwD; ii) explore whether the health benefits of EXCITE-PAC, if any, are mediated through improved PAC at the 36-week (i.e., about 6 months) follow-up endpoints; and iii) explore carers' perceptions of the benefits, limitations and acceptability of the EXCITE-PAC programme.

Objectives i) To evaluate the effects of the existential-cognitive intervention to enhance the positive aspects of caregiving (EXCITE-PAC) on PAC and the health outcomes of family carers of persons living with dementia (PLwD).

ii) To evaluate whether the positive health effects of EXCITE-PAC, if any, are mediated through a change in PAC.

iii) To explore the experience of family carers in engaging with EXCITE-PAC, as well as the perceived intervention effects.

Hypotheses

Family carers who receive the 12-week EXCITE-PAC programme will report more positive changes in i) PAC, ii) HRQoL, iii) depression, iv) self-efficacy in caregiving, and v) meaning-making upon programme completion (12 weeks), and at 24 weeks and 36 weeks, than those who receive a 12-week education programme on dementia caregiving.

The changes in HRQoL and depression among family carers from baseline to the three post-test endpoints will be mediated by an improvement in PAC.

Research method

1. Study setting and participants

   This sequential mixed-method study will include a double-blind randomised controlled trial and a post-trial qualitative study. Blinding procedures will be achieved in that the data collectors for the post-test results will be blinded to group status, and participants will not be informed about whether EXCITE-PAC or structured education is the tested intervention. They will only be informed that they have been assigned to Programme A or Programme B. Family carers of PLwD will be recruited from dementia caregiver hubs supported by various NGOs. The inclusion criteria are: i) family carers of Chinese PLwD diagnosed at least six months previously; ii) caregiving for ≥ 4 hours/day; iii) Chinese-speaking; iv) having a mobile device to access virtual meetings via GoToMeeting or Zoom; and v) providing consent to participate. Power analysis guides the sample size estimation. Although no study to date has adopted the existential positive psychology paradigm to improve PAC, a systematic review reported the effect size (Hedges' g) of a non-pharmacological intervention on PAC to be 0.31 and 0.89 for the post-intervention and follow-up evaluations, respectively, with the inclusion of counselling or psychotherapy further enhancing the effect. The investigators thus conservatively assume that EXCITE-PAC will achieve at least a small effect of 0.35 on PAC. A total of 304 family carers will be needed (power: 80%; α: 0.05; attrition rate: 15%). Permuted block randomisation (block size: 8, 12, 16) with computer-generated random codes will be performed to allocate participants in a 1:1 ratio to the EXCITE-PAC or education programme using the "sequentially numbered, opaque sealed envelopes" procedure. This sample size is sufficient to conduct path analysis examining the mediating effects of PAC.

   For the qualitative interviews, a purposive subsample of 30 family carers who have completed the EXCITE-PAC programme will be recruited. To optimise sample variation, participants with different treatment responses to EXCITE-PAC will be recruited, with 10 participants each from the 0-35th percentile, >35th-70th percentile and >70th percentile ranges of change in PAC, and variation in the sample's socio-demographic characteristics will also be maximised. The interviews will be audio-recorded for analysis.
2. Tested intervention: EXCITE-PAC

The 12-week EXCITE-PAC programme is underpinned by existential positive psychology, which integrates the use of self-distancing cognitive reappraisal techniques to enhance emotional regulation and meaning-making with respect to the purpose and significance of dementia caregiving. A strength-based approach that includes narrative and empowerment strategies will be integrated to further optimise meaning-making in the dimensions of sense of coherence (SOC) and self-efficacy in caregiving. A research assistant (RA1) with a Bachelor's degree in psychology, gerontology or social science will deliver the intervention. The multi-disciplinary research team, which has expertise in cognitive-behavioural, narrative and empowerment interventions, and dementia caregiving, will provide two weeks of training. A standard protocol has been developed to guide the implementation of EXCITE-PAC, the overall design of which is outlined in Figure 2.

The 12-week EXCITE-PAC programme adopts a hybrid mode, including a face-to-face home visit (Week 1), group-based virtual meetings (Weeks 2-8), and telephone follow-ups (Weeks 10-12). EXCITE-PAC will commence with a home visit to establish narrative-based caregiver biographies. Over the next seven weeks, weekly virtual group-based meetings will be held, during which video-guided self-distancing cognitive reappraisal will be used to enhance emotional regulation and meaning-making. The goal-oriented empowerment approach will be used in the virtual meetings to facilitate carers' use of reframing and refocusing techniques in the day-to-day caregiving process to promote the PAC. Thereafter, two bi-weekly telephone calls will be made to continue supporting goal attainment. The details of EXCITE-PAC are as follows.

Narrative-based caregiver biographies (face-to-face home visit) EXCITE-PAC will commence by establishing each carer's caregiving biography using narrative strategies. The purpose is to engage caregivers in reflection on the caregiving journey, particularly on their initial motivation to engage in caregiving, their relationship with the PLwD since the premorbid stage, and how they have coped with caregiving hardships and challenges in the past. With reference to the predictive model of PAC, carers' reflection on their initial motivation and relationship will set a context favourable to PAC evolvement through emotional regulation. Increasing their awareness of past successes can also help to improve their SOC, which is an important dimension in the meaning-making of the experience of dementia caregiving.

The caregiving biography is a tailored booklet to document the caregiving journey, with the content discussed during the home visit (i.e., motivation to care, relationship with PLwD, ways to overcome hardship in the past and personal strengths). Narrative strategies, including externalising and re-authoring conversations, will be used to enhance disclosure. The externalising conversation strategy is based on the assumption that people who internalise a persistent problem have a delimited view of the problematic issue. To externalise the challenging caregiving situation, the biography will use 'life adventure' as a metaphor for the caregiving journey. The carers will be guided to describe how and why their caregiving role commenced and how their relationship with the PLwD has evolved. Stickers with different descriptors will be provided to facilitate the process, and carers will be asked to elaborate on why a particular sticker has been chosen. To direct their attention to previous performance successes, they will be asked to mark and label their most challenging time on the trail with a place (e.g., desert, tunnel), and to describe how they left the place (i.e., overcame the hardship). Their current caregiving challenges will also be explored. Re-authoring questions will be used to deliberately identify exceptions to problem-saturated caregiving (i.e., exceptional success in managing a challenging caregiving situation). The interveners will conduct situation analysis with the caregivers to identify the factors (e.g., actions, events and personal strengths or characteristics) leading to such exceptional situations. Their responses will help the interveners to identify and highlight the generalised resistance resources (GRRs) from the internal and external environments of carers. In this way, the carers will be better able to recognise their own personal strengths to tackle challenging caregiving situations. The completed biographies will be kept by the carers.

Self-distancing reappraisal for cognitive emotional regulation (2nd-5th virtual meetings) These group-based sessions will be delivered via GoToMeeting with the aim of capitalising on the carers' abilities to engage in cognitive emotional regulation. Each group will have 3-4 carers to enhance peer sharing. Each of the four sessions will cover emotional regulation in relation to: i) handling cognitive decline and functional dependence; ii) BPSD and social interaction with PLwD; iii) family dynamics; and iv) caregiving role demands. The impact of emotional arousal on caregiving role adaptation will be explained at the outset. Self-distancing reappraisal will be used by displaying a micro-movie to illustrate the thought-emotion-behaviour relationship relevant to the session topic. The micro-movies were developed based on reflective notes capturing the dementia caregiving experience in our previous GRF project. The carers will be guided to identify the thought-emotion-behaviour relationship in the scenario presented. They will then be invited to share similar encounters, with the focus placed on exploring their emotional manifestation in that episode (i.e., how and why) and discussing how such emotions affect their role perception, relationship with PLwD and overall well-being. Next, a micro-movie demonstrating how a change in thought processes in the same scenario can prevent negative emotional arousal will be shared. A 5-step empowerment approach will be used in each session to engage carers in setting goal-oriented action plans to enhance emotional regulation. The goal and action plan will be documented in the carer biographies for follow-up in the next session.

Self-distancing reappraisal for meaning-making (6th-8th virtual meetings) These group sessions aim to use cognitive reappraisal strategies to engage the caregivers in meaning-making. Although meaning-making is a person-centred process, a group format will be adopted, as our previous study demonstrated the positive peer influence on widening the life space and opportunities of carers and supporting each other to more positively construe role adaptation.24 Our review suggests that meaning-making contributes to the PAC domains: mutuality in the dyadic relationship, family cohesion and functionality, and personal growth and purpose in life. These three sessions will hence focus on these areas. Each session will commence with a micro-movie demonstrating a 4-stop caregiving journey: 1) the pre-morbid situation, 2) the changes imposed by caregiving, 3) how carers adjust and 4) how they develop new meaning from the situation. Each movie will cover the evidence the investigators identified for each PAC domain. Then, the carers will be invited to share their own situations using the 4-stop journey as outlined in the movie. An accepting atmosphere will be adopted to invite negative responses. Peers will be invited to provide their perspectives to support meaning-making. The identified meanings will be documented in the biographies to enhance reflection and retention.

Telephone follow-up (Weeks 9-12) Two telephone follow-up calls will be made to carers to follow up on goal attainment and reinforce their strengths, emotional regulation, and new meaning-making.

ELIGIBILITY:
Inclusion Criteria:

* family carers of Chinese PLwDs diagnosed at least six months previously
* caregiving for ≥ 4 hours/day
* Chinese-speaking
* have a mobile device to access virtual meeting via Go-To-Meeting or Zoom
* consent to participate

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The Positive Aspect of Caregiving Instrument | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate self-affirmation and outlook on life. It is a 5-point Likert scale, with higher total scores (ranging from 11-55) indicating a more positive perception of the caregiving role.
The Caregiving Self-Efficacy Scale | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate self-efficacy of carers in managing disturbing behaviour, controlling upsetting thoughts and obtaining a respite in caring for of the PLwD, with higher scores representing greater self-confidence. It is a 15-item tool used to assess caregivers' confidence in managing caregiving situations, rated on a 0-100 scale. Higher score indicate stronger self-efficacy.
The Meaning-Focused Coping Scale | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate meaning-focused coping, including changes in situational and global beliefs, goals, meaning making, long-term prevention strategies, rational resource use, acceptance and heuristic thinking. It is a 26-items tool using a 7-point Likert scale, higher scores indicating a higher level of meaning-focused coping.
The 10-item Centre of Epidemiological Studies Depression Scale | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate affective symptoms reflecting depression on an ascending 4-point scale of increasing severity.

SECONDARY OUTCOMES:
The Medical Outcomes Study Short Form Health Survey | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate the quality of life with 8 dimensional scores and two component scores to capture physical and mental health. Higher scores indicate less disability
Positive Affect Index | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate the participants' positive affect toward the dementia patient. The higher score indicate higher positive affect of respondant.
The Intrinsic Motivations to Care | Baseline (T0), Up to 12 weeks (T1), up to 24 weeks (T2), up to 36 weeks (T3).
  To evaluate the intrinsic motivations of family caregivers to provide care to the PWD. The scale generally uses a 7-point Likert scale (ranging from 1, "not at all true" to 7, "very true") to gauge the intensity of motivation.

CONTACTS AND LOCATIONS:
Overall Officials: YU YU, RN, PhD, FHKAN, FAAN, FGSA, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Younas A, Pedersen M, Durante A. Characteristics of joint displays illustrating data integration in mixed-methods nursing studies. Journal of Advanced Nursing, 2020. 76(2): 676-686.
- [Background] Elo, S., & Kyngäs, H. The qualitative content analysis process. Journal of Advanced Nursing, 2008, 62(1):107-115.
- [Background] Preacher, K. J., & Hayes, A. F. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behavior Research Methods, 2008, 40(3): 879-891.
- [Background] Hu, L., & Bentler, P. Cutoff criteria for fit indexes in covariance structure analysis: Conventional criteria versus new alternatives. Structural Equation Modeling: A Multidisciplinary Journal, 1999, 6(1): 1-55.
- [Background] Rosseel Y; lavaan: An R Package for Structural Equation Modeling. Journal of Statistical Software 2012;48(2):1 - 36. doi: 10.18637/jss.v048.i02.
- [Background] Singer JD, Willett JB. Applied longitudinal data analysis: modelling change and event occurrence. New York: Oxford University Press, 2003.
- [Background] Lyonette, C., & Yardley, L. The influence on carer wellbeing of motivations to care for older people and the relationship with the care recipient. Ageing and Society, 2003, 23(4), 487-506.
- [Background] Quinn C, Clare L, Woods RT. What predicts whether caregivers of people with dementia find meaning in their role? International Journal of Geriatric Psychiatry 2012; 27:1195-1202.
- [Background] Bengston, V, Schrader, S. Parent-child relations. In Mangen DJ, Peterson WA (eds.), Research Instruments in Social Gerontology (pp. 115-185). Minneapolis, MN: University of Minneapolis Press, 1982.
- [Background] Leung VP, Lam LC, Chiu HF, Cummings JL, Chen QL. Validation study of the Chinese version of the neuropsychiatric inventory. International Journal of Geriatric Psychiatry, 2000, 16(8):789-93.
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 Health Survey valid and equivalent for a Chinese population? Quality of Life Research. 2005, 4:539-547.
- [Background] Amirkhan, J., & Greaves, H. Sense of Coherence and Stress: The Mechanics of a Healthy Disposition. Psychology & Health, 2003, 18(1): 31-62. https://doi.org/10.1080/0887044021000044233
- [Background] Cheng, S., & Chan, A. The Center for Epidemiologic Studies Depression Scale in older Chinese: Thresholds for long and short forms. International Journal of Geriatric Psychiatry, 2005, 20(5): 465-470.
- [Background] Gan Y, Guo M, Tong J. Scale development of meaning-focused coping. Journal of Loss and Trauma, 2013; 18: 10-26.
- [Background] Au A, Lai M, Lau K, Pan P, Lam L. Social support and well-being in dementia family caregivers.: the mediating role of self-efficacy. Aging & Mental Health 2009, 3:761-768.
- [Background] Lou VWQ, Lau BHP, Cheung KSL. Positive aspects of caregiving: Scale validation among Chinese dementia caregivers (CG). Achieves of Gerontology & Geriatrics 2015, 60: 299-306.
- [Background] Yu DSF, Cheng ST, Wang J. Unravelling positive aspects of caregiving in dementia: An integrative review of research literature. International Jouranl of Nursing Studies. 2018 Mar;79:1-26.
- [Background] Yu DSF, Cheng ST, Chow EOW, Kwok T, McCormack B, Wu W. The effects of a salutogenic strength-based intervention on sense of coherence and health outcomes of dementia family carers: A randomized controlled trial, Age and Ageing, 2023, 52(9): afad160
- [Background] Loehlin, John C. Latent Variable Models: An Introduction to Factor, Path, and Structural Equation Analysis (4th ed.). Psychology Press, 2004.
- [Background] Park CL. The Meaning Making Model: A framework for understanding meaning, spirituality, and stress-related growth in health psychology. The Eur Health Psychologist, 2013; 15: 40-47.
- [Background] Hedeker, D., Gibbons, R., & Waternaux, C. Sample Size Estimation for Longitudinal Designs with Attrition: Comparing Time-Related Contrasts between Two Groups. Journal of Educational and Behavioural Statistics, 1999, 24(1): 70-93.
- [Background] Cheng ST, Li KK, Losada A, Zhang F, Au A, Thompson LW, Gallagher-Thompson D. The effectiveness of nonpharmacological interventions for informal dementia caregivers: An updated systematic review and meta-analysis. Psychology and Aging, 2020, 35(1):55-77.
- [Background] Mittelmark MB, Bauer GF. Salutogenesis as a Theory, as an Orientation and as the Sense of Coherence. 2022 Jan 1. In: Mittelmark MB, Bauer GF, Vaandrager L, et al., editors. The Handbook of Salutogenesis [Internet]. 2nd edition. Cham (CH): Springer; 2022.
- [Background] Tropen Y, Liberman N. "Construal-level theory of psychological distance". Psychological Review. 2010, 117 (2): 440-463.
- [Background] González-Prendes, A., & Resko, S. M. (2012). Cognitive-behavioral theory. Trauma: Contemporary directions in theory, practice, and research, 14-41.
- [Background] Wong PT P. Existential positive psychology. In S. Lopez (Ed.), Encyclopedia of positive psychology (2nd ed.). Oxford, UK: Wiley Blackwell
- [Background] Yu DSF, Cheng ST, Chen K, Predicting positive aspect of caregiving in a dementia caregiving context: a longitudinal model testing. International Journal of Nursing Studies. Under review.
- [Background] Yu DSF, Cheng ST, Kwok T. Developing and testing of an integrative theoretical model to predict positive aspects of caregiving among family caregivers of persons with dementia: A study protocol. Journal of Advanced Nursing. 2021 Jan;77(1):401-410.
- [Background] Mausbach BT, Coon DW, Depp C, Rabinowitz YG, Wilson-Arias E, Kraemer HC, Thompson LW, Lane G, Gallagher-Thompson D. Ethnicity and time to institutionalization of dementia patients: a comparison of Latina and Caucasian female family caregivers. Journal of American Geriatric Society 2004; 52:1077-1084.
- [Background] Hirschfeld M. Home care versus institutionalization: family caregiving and senile brain disease. Int J Nurs Stud 2003; 40:463-469.
- [Background] Cohen CA, Gold DP, Shulman KI, Zucchero CA. Positive aspects in caregiving: An overlooked variable in research. Canadian Journal of Aging 1994; 13:378-391.
- [Background] Rapp SR, Chao D. Appraisals of strain and of gain: Effects on psychological wellbeing of caregivers of dementia patients. Aging and Mental Health 2000; 4:142-147.
- [Background] Williams IC. Emotional health of black and white dementia caregivers: A contextual examination. J Gerontol B Psychol Sci Soc Sci 2005; 60: P287-P295.
- [Background] Narayan S, Lewis M, Tornatore J, Hepburn K, Corcoran-Perry S. Subjective responses to caregiving for a spouse with dementia. Journal of Gerontological Nursing 2001; 27:19-28.
- [Background] Andrén S, Elmståhl S. Family caregivers' subjective experiences of satisfaction in dementia care: aspects of burden, subjective health and sense of coherence. Scandinavian Journal of Caring Science 2005; 19:157-168.
- [Background] Valimaki T.H., Martikainen J.A., Hongisto K., Vaatainen S., Sintonen H., Koivisto A.M. Impact of Alzheimer's disease on the family caregiver's long-term quality of life: Results from an ALSOVA follow-up study. Qual. Life Res. 2016;25:687-697.
- [Background] Shin JH, Kim JH. Family Caregivers of People with Dementia Associate with Poor Health-Related Quality of Life: A Nationwide Population-Based Study. International Journal of Environmental Research and Public Health. 2022 Dec 5;19(23):16252.
- [Background] Papastavrou E, Kaloderinou A, Papacostas SS, Tsangari H, Sourtzi P. Caring for a relative with dementia: Family caregiver burden. Journal of Advanced Nursing 2007; 58: 446-457.
- [Background] Global action plan on the public health response to dementia 2017-2025. Geneva: World Health Organization; 2017. License: CC BY-NC-SA 3.0 IGO.
- [Background] Alzhimer disease international. Dementia statistics. Access from https://www.alzint.org/about/dementia-facts-figures/dementia-statistics/ on 27th Sept 2023